CLINICAL TRIAL: NCT02898779
Title: Development of Safer Drugs for Malaria in U.S. Troops, Civilian Personnel, and Travelers: Clinical Evaluation of Primaquine Enantiomer
Brief Title: Metabolism and Pharmacokinetics of Primaquine Enantiomers in Human Volunteers, Study 1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Mississippi, Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: PQ Study 1
Record Dates: First submitted 2016-07-21; First posted 2016-09-13 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — Primaquine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 ( Primaquine Low Dose) (Experimental): Interventions: Primaquine, R-Primaquine, S-Primaquine, SR Primaquine A single center, prospective, cross-over, randomized phase 1 trial. Thirty-six participants, enrolled into a two cohort pharmacokinetic study evaluating two dose levels of primaquine isomers.
  Cohort 1 (Low Dose Level)- single dose of 15 mg of S-Primaquine and 15 mg of R-Primaquine compared to 30 mg RS-Primaquine over 24 hours. Participants will cross-over after a one week wash-out period.
  Interventions: Drug: Primaquine, R-Primaquine, S-Primaquine, SR Primaquine
- Cohort 2 (Primaquine High Dose) (Experimental): Interventions: Primaquine, R-Primaquine, S-Primaquine, SR Primaquine A single center, prospective, cross-over, randomized phase 1 trial. Thirty-six participants, enrolled into a two cohort pharmacokinetic study evaluating two dose levels of primaquine isomers.
  Cohort 2 (High Dose Level)-single dose of 22.5 mg of S-Primaquine and 22.5 mg of R-Primaquine compared to 45 mg RS-Primaquine over 24 hours. Participants will cross-over among the treatment arms following a one week wash-out period between each.
  Interventions: Drug: Primaquine, R-Primaquine, S-Primaquine, SR Primaquine

INTERVENTIONS:
Drug: Primaquine, R-Primaquine, S-Primaquine, SR Primaquine — Cohort 1: Eighteen individuals (6 per group) Cohort 2: Eighteen individuals (6 per group)
  Group 1-15 mg of S-Primaquine followed by one-week washout, 15 mg of R-Primaquine followed by one week washout, and 30 mg of RS-Primaquine.
  Group 2- 15 mg of R-Primaquine followed by one-week washout, 30 mg of RSPQ followed by one week washout, and 15 mg of SPQ.
  Group 3- 30 mg of RS-Primaquine followed by one week washout,15 mg of SPQ followed by a one week washout, and 15 mg of RPQ.
  Other Names: Primaquine

SUMMARY:
To investigate the comparative tolerability, metabolism and pharmacokinetics of individual enantiomers of PQ in healthy human volunteers. The specific aim is the comparative evaluation of the metabolism, pharmacokinetic behavior, and tolerability of the isomers of PQ (RPQ and SPQ and the racemic mixture RSPQ) in normal healthy human volunteers.

DETAILED DESCRIPTION:
The primary objective of this project is to investigate the comparative tolerability, metabolism and pharmacokinetics of individual enantiomers of PQ in healthy human volunteers.

The overall approach is as follows: in 36 healthy volunteers with documented normal G6PD activity, we will administer a single oral dose of RPQ, SPQ, or RSPQ. At various times after dosing, we will draw blood samples, in which we will record the plasma levels of the parent drugs, along with plasma and urinary metabolites. The comparative pharmacokinetics, tolerability and hematological effects of these two enantiomers and the racemate will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18-60 years of age)
* Informed consent
* Healthy

Exclusion Criteria:

* Known history of liver, kidney or hematological disease;
* known history of cardiac disease, arrhythmia, QT prolongation;
* Autoimmune disorder;
* Report of an active infection;
* Evidence of G6PD deficiency

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Primary outcome: Plasma concentration of parent primaquine and carboyprimaquine following a single dose treatment with primaquine (racemate or enantiomers) not to exceed 45 mg | between 0-24 Hours
  This study would provide information on differential pharmacokinetics and metabolism of enantiomers of primaquine in normal human volunteers

SECONDARY OUTCOMES:
Area Under Curve (AUC) for primaquine up to 24 hours after the primaquine administration | between 0-24 hours
  This study would provide information on differential pharmacokinetics and metabolism of enantiomers of primaquine in normal human volunteers
Maximum concentration (Cmax) for primaquine up to 24 hours after the primaquine administration | between 0-24 hours
  This study would provide information on differential pharmacokinetics and metabolism of enantiomers of primaquine in normal human volunteers
Area Under Curve (AUC) for carboxyprimaquine, the major plasma metabolite of primaquine, up to 24 hours after primaquine administration | between 0-24 hours
  This study would provide information on differential pharmacokinetics and metabolism of enantiomers of primaquine in normal human volunteers
Maximum concentration of carboxyprimaquine, the major plasma metabolite of primaquine, up to 24 hours after primaquine administration | between 0-24 hours
  This study would provide information on differential pharmacokinetics and metabolism of enantiomers of primaquine in normal human volunteers
Maximum concentration of selected metabolites primaquine (other than carboxyprimaquine) up to 24 hours after primaquine administration | between 0-24 hours
  This study would provide information on differential pharmacokinetics and metabolism of enantiomers of primaquine in normal human volunteers. The exact nature of these metabolites will be determined from previous animal and human studies
hemoglobin and methemoglobin levels in the blood after administration of primaquine | 0-72 hours
  To monitor hemoglobin and methemoglobin levels in normal human volunteers treated with single dose of primaquine not to exceed 45 mg
Genotyping of Cytochrome P-450 (CYP) | day 0
  To determine correlation between metabolism of primaquine and CYP 2D6 genotype

CONTACTS AND LOCATIONS:
Overall Officials: Babu L Tekwani, Ph.D, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi, Oxford, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Avula B, Tekwani BL, Chaurasiya ND, Nanayakkara NP, Wang YH, Khan SI, Adelli VR, Sahu R, Elsohly MA, McChesney JD, Khan IA, Walker LA. Profiling primaquine metabolites in primary human hepatocytes using UHPLC-QTOF-MS with 13C stable isotope labeling. J Mass Spectrom. 2013 Feb;48(2):276-85. doi: 10.1002/jms.3122. PMID 23378100
- [Result] Avula B, Khan SI, Tekwani BL, Nanayakkara NP, McChesney JD, Walker LA, Khan IA. Analysis of primaquine and its metabolite carboxyprimaquine in biological samples: enantiomeric separation, method validation and quantification. Biomed Chromatogr. 2011 Sep;25(9):1010-7. doi: 10.1002/bmc.1557. Epub 2010 Nov 5. PMID 21058417
- [Result] Baker JK, McChesney JD. Differential metabolism of the enantiomers of primaquine. J Pharm Sci. 1988 May;77(5):380-2. doi: 10.1002/jps.2600770503. PMID 3411455
- [Result] Lu H. Stereoselectivity in drug metabolism. Expert Opin Drug Metab Toxicol. 2007 Apr;3(2):149-58. doi: 10.1517/17425255.3.2.149. PMID 17428147
- [Result] Fasinu PS, Tekwani BL, Nanayakkara NP, Avula B, Herath HM, Wang YH, Adelli VR, Elsohly MA, Khan SI, Khan IA, Pybus BS, Marcsisin SR, Reichard GA, McChesney JD, Walker LA. Enantioselective metabolism of primaquine by human CYP2D6. Malar J. 2014 Dec 17;13:507. doi: 10.1186/1475-2875-13-507. PMID 25518709
- [Result] Fasinu PS, Avula B, Tekwani BL, Nanayakkara NP, Wang YH, Bandara Herath HM, McChesney JD, Reichard GA, Marcsisin SR, Elsohly MA, Khan SI, Khan IA, Walker LA. Differential kinetic profiles and metabolism of primaquine enantiomers by human hepatocytes. Malar J. 2016 Apr 19;15:224. doi: 10.1186/s12936-016-1270-1. PMID 27093859
- [Result] Graves PM, Gelband H, Garner P. Primaquine or other 8-aminoquinoline for reducing Plasmodium falciparum transmission. Cochrane Database Syst Rev. 2015 Feb 19;(2):CD008152. doi: 10.1002/14651858.CD008152.pub4. PMID 25693791
- [Result] Jin X, Pybus BS, Marcsisin R, Logan T, Luong TL, Sousa J, Matlock N, Collazo V, Asher C, Carroll D, Olmeda R, Walker LA, Kozar MP, Melendez V. An LC-MS based study of the metabolic profile of primaquine, an 8-aminoquinoline antiparasitic drug, with an in vitro primary human hepatocyte culture model. Eur J Drug Metab Pharmacokinet. 2014 Jun;39(2):139-46. doi: 10.1007/s13318-013-0139-8. PMID 23797843
- [Result] Mihaly GW, Ward SA, Edwards G, Orme ML, Breckenridge AM. Pharmacokinetics of primaquine in man: identification of the carboxylic acid derivative as a major plasma metabolite. Br J Clin Pharmacol. 1984 Apr;17(4):441-6. doi: 10.1111/j.1365-2125.1984.tb02369.x. PMID 6721990
- [Result] Nanayakkara NP, Ager AL Jr, Bartlett MS, Yardley V, Croft SL, Khan IA, McChesney JD, Walker LA. Antiparasitic activities and toxicities of individual enantiomers of the 8-aminoquinoline 8-[(4-amino-1-methylbutyl)amino]-6-methoxy-4-methyl-5-[3,4-dichlorophenoxy]quinoline succinate. Antimicrob Agents Chemother. 2008 Jun;52(6):2130-7. doi: 10.1128/AAC.00645-07. Epub 2008 Mar 31. PMID 18378716
- [Result] Nanayakkara NP, Tekwani BL, Herath HM, Sahu R, Gettayacamin M, Tungtaeng A, van Gessel Y, Baresel P, Wickham KS, Bartlett MS, Fronczek FR, Melendez V, Ohrt C, Reichard GA, McChesney JD, Rochford R, Walker LA. Scalable preparation and differential pharmacologic and toxicologic profiles of primaquine enantiomers. Antimicrob Agents Chemother. 2014 Aug;58(8):4737-44. doi: 10.1128/AAC.02674-13. Epub 2014 Jun 9. PMID 24913163
- [Result] Potter BM, Xie LH, Vuong C, Zhang J, Zhang P, Duan D, Luong TL, Bandara Herath HM, Dhammika Nanayakkara NP, Tekwani BL, Walker LA, Nolan CK, Sciotti RJ, Zottig VE, Smith PL, Paris RM, Read LT, Li Q, Pybus BS, Sousa JC, Reichard GA, Marcsisin SR. Differential CYP 2D6 metabolism alters primaquine pharmacokinetics. Antimicrob Agents Chemother. 2015 Apr;59(4):2380-7. doi: 10.1128/AAC.00015-15. Epub 2015 Feb 2. PMID 25645856
- [Result] Pybus BS, Marcsisin SR, Jin X, Deye G, Sousa JC, Li Q, Caridha D, Zeng Q, Reichard GA, Ockenhouse C, Bennett J, Walker LA, Ohrt C, Melendez V. The metabolism of primaquine to its active metabolite is dependent on CYP 2D6. Malar J. 2013 Jun 20;12:212. doi: 10.1186/1475-2875-12-212. PMID 23782898
- [Result] Saunders D, Vanachayangkul P, Imerbsin R, Khemawoot P, Siripokasupkul R, Tekwani BL, Sampath A, Nanayakkara NP, Ohrt C, Lanteri C, Gettyacamin M, Teja-Isavadharm P, Walker L. Pharmacokinetics and pharmacodynamics of (+)-primaquine and (-)-primaquine enantiomers in rhesus macaques (Macaca mulatta). Antimicrob Agents Chemother. 2014 Dec;58(12):7283-91. doi: 10.1128/AAC.02576-13. Epub 2014 Sep 29. PMID 25267666
- [Result] Schmidt LH, Alexander S, Allen L, Rasco J. Comparison of the curative antimalarial activities and toxicities of primaquine and its d and l isomers. Antimicrob Agents Chemother. 1977 Jul;12(1):51-60. doi: 10.1128/AAC.12.1.51. PMID 407841
- [Result] Tekwani BL, Walker LA. 8-Aminoquinolines: future role as antiprotozoal drugs. Curr Opin Infect Dis. 2006 Dec;19(6):623-31. doi: 10.1097/QCO.0b013e328010b848. PMID 17075340
- [Result] Tekwani BL, Avula B, Sahu R, Chaurasiya ND, Khan SI, Jain S, Fasinu PS, Herath HM, Stanford D, Nanayakkara NP, McChesney JD, Yates TW, ElSohly MA, Khan IA, Walker LA. Enantioselective pharmacokinetics of primaquine in healthy human volunteers. Drug Metab Dispos. 2015 Apr;43(4):571-7. doi: 10.1124/dmd.114.061127. Epub 2015 Jan 30. PMID 25637634
- [Result] Vale N, Moreira R, Gomes P. Primaquine revisited six decades after its discovery. Eur J Med Chem. 2009 Mar;44(3):937-53. doi: 10.1016/j.ejmech.2008.08.011. Epub 2008 Sep 11. PMID 18930565
- [Result] Vasquez-Vivar J, Augusto O. Hydroxylated metabolites of the antimalarial drug primaquine. Oxidation and redox cycling. J Biol Chem. 1992 Apr 5;267(10):6848-54. PMID 1313024